CLINICAL TRIAL: NCT02916862
Title: Effect of Soluble Corn Fiber Supplementation for 1 Year on Bone Metabolism in Adolescents
Acronym: MetA-Bone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Cristina Palacios, PhD, Professor and Chair, Florida International University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 107593; 1R01HD098589-01 (NIH)
Record Dates: First submitted 2016-08-25; First posted 2016-09-28 (Estimated); Results first posted 2025-10-29 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Osteoporosis
Keywords: fiber; calcium absorption; bone mass; adolescents
MeSH Terms: conditions — Osteoporosis | interventions — Calcium

STUDY DESIGN:
Intervention Model Description: we are testing a fiber and calcium supplement so it is not a drug
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Soluble Corn Fiber (SCF) + Calcium (Experimental): This group will receive 12 g/d of soluble corn fiber (SCF) + 600 mg/d of elemental calcium carbonate, administered twice a day
  Interventions: Combination Product: Soluble Corn Fiber (SCF) + Calcium
- Soluble Corn Fiber (SCF) without calcium (Active Comparator): This group will receive 12 g/d of soluble corn fiber (SCF) + 600 mg/d of elemental calcium carbonate, administered twice a day
  Interventions: Dietary Supplement: Soluble Corn Fiber (SCF) without Calcium
- Placebo (Placebo Comparator): This group will receive a similar supplement without SCF or calcium, administered twice a day
  Interventions: Dietary Supplement: Placebo
- Placebo + calcium (Placebo Comparator): This group will receive a similar supplement without SCF + 600 mg/d of elemental calcium carbonate, administered twice a day
  Interventions: Combination Product: Placebo + calcium

INTERVENTIONS:
Dietary Supplement: Soluble Corn Fiber (SCF) without Calcium — Participants will consume a supplement with 12 g/day of SCF for 12 months
  Arms: Soluble Corn Fiber (SCF) without calcium
Combination Product: Soluble Corn Fiber (SCF) + Calcium — Participants will consume a supplement with 12 g/day of SCF + calcium carbonate (600 mg/day) for 12 months
  Arms: Soluble Corn Fiber (SCF) + Calcium
Dietary Supplement: Placebo — Participants will consume a supplement without SCF or calcium carbonate for 12 months
  Arms: Placebo
Combination Product: Placebo + calcium — Participants will consume a supplement without SCF + calcium carbonate (600 mg/day) for 12 months
  Arms: Placebo + calcium

SUMMARY:
The primary aim of this proposal is to determine the effects of soluble corn fiber (SCF) supplementation for 1 year on bone metabolism in growing adolescents compared to controls. For the proposed study, a randomized double-blinded placebo controlled clinical trial will be conducted in 236 healthy adolescents aged 10-13 years, equally randomly assigned to one of four intervention groups: SCF (12 g/d), SCF + calcium (12 g/d of SCF + 600 mg/d of elemental calcium), placebo (0 g/d of SCF or of calcium), and placebo + calcium (0 g/d of SCF + 600 mg/d of elemental calcium); all administered twice a day. Bone mass will be assessed at baseline at 6 months and at 12 months and bone related biomarkers and fecal microbiome will be assessed at baseline and at 12 months.

DETAILED DESCRIPTION:
The adolescent period is crucial for optimizing future bone health because bone accumulates rapidly during these years and accounts for up to half of adult peak bone mass. Calcium intake during this period is critical for adequate bone mineralization but this is the nutrient most deficient in the diets of adolescents. A strategy to maximize bone mineralization during this critical period is to increase the absorption of the calcium being consumed. This could be achieved by supplementing diets with certain non-digestible carbohydrates, such as soluble corn fiber (SCF).

The primary aim of this study is to determine the effects of SCF supplementation for 1 year on bone metabolism in growing adolescents compared to controls. A randomized double-blinded placebo controlled clinical trial will be conducted in 236 healthy adolescents aged 10-13 years, equally randomly assigned to one of four intervention groups: SCF (12 g/d), SCF + calcium (12 g/d of SCF + 600 mg/d of elemental calcium), placebo (0 g/d of SCF or of calcium), and placebo + calcium (0 g/d of SCF + 600 mg/d of elemental calcium); all administered twice a day. Bone mass will be assessed at baseline at 6 months and at 12 months and bone related biomarkers and fecal microbiome will be assessed at baseline and at 12 months. The treatments will be provided in the form of flavored drinks twice per day (this was previously used in a short-term study among adolescents with excellent acceptance). Bone mass and anthropometric measurements will be assessed at baseline, at 6 months and at 12 months and bone related biomarkers and fecal microbiome will be assessed at baseline and at 12 months. Assessment visits will be conducted in the Clinical Research Center of the Stempel School of Public Health at Florida International University. We will also have short home visits at 3 and 9 months to collect unused supplements and provide more supplements. In all visits, participants will complete several questionnaires, such as general health, diet and activity questionnaire. Compliance will be evaluated at all visits and also in real time using a study mobile app.

The primary outcome is change in bone mineral content (BMC) measured using Dual-energy X-ray absorptiometry (DXA)

The secondary outcomes include biochemical markers reflecting vitamin D status, calcium homeostasis and bone, such as serum calcium, phosphorus, creatinine, osteocalcin, carboxy-terminal collagen crosslinks (CTX), parathyroid hormone (PTH), bone specific alkaline phosphatase, 25-(OH) vitamin D3, 1,25-(OH)2 vitamin D3, and insulin growth factor 1 (IGF-I) and urinary calcium, phosphorus, creatinine and N-telopeptide cross-links.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between the 5th and 85th percentiles for age and sex based on the Centers for Disease Control Growth Charts.

Exclusion Criteria:

* Subjects with any chronic illness requiring regular medication use.
* Those taking calcium supplements (>500 mg/d) and vitamin D supplements (>400 IU/d) on a regular basis

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 177 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Palacios, PhD, Principal Investigator — Department of Dietetics, College of Public Health, Florida International Univ.
Locations (1):
- Flroida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators outside the research team will only be granted access to the data after their proposal has been evaluated and approved by the research team and by the Florida International University Office of Research Integrity. We will only provide access to the samples and de-identified data as required to address the proposed research goals and only under a data-sharing agreement.
Supporting Information: Study Protocol, ICF
Time Frame: When the primary outcome is completed.
Access Criteria: We will share the data and associated documentation only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Derived] Palacios C, Leone J, Clayton P, Hernandez J, Trak-Fellermeier MA, Macchi A, Ramirez-Roggio D, Cobo Y, Bautista S, Connelly J, Elington M, Romero J, Galvan R. Effectiveness and costs of the recruitment strategies used in the MetA-Bone trial, a randomized clinical trial to test the effects of soluble corn fiber supplementation for 1 year in children. Contemp Clin Trials. 2024 Dec;147:107715. doi: 10.1016/j.cct.2024.107715. Epub 2024 Oct 15. PMID 39413989

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Although 213 were recruited (signed consent form), only 177 completed the randomization visit and were randomized.
Pre-assignment Details: Randomization was pre-determined using a block randomization document, which was computer generated.
Groups:
- Soluble Corn Fiber (SCF) + Calcium: This group received 12 g/d of soluble corn fiber (SCF) + 600 mg/d of elemental calcium carbonate, administered twice a day
  Soluble Corn Fiber (SCF) + Calcium: Participants consumed a supplement with 12 g/day of SCF + calcium carbonate (600 mg/day) for 12 months
- Soluble Corn Fiber (SCF) Without Calcium: This group received 12 g/d of soluble corn fiber (SCF) + 600 mg/d of elemental calcium carbonate, administered twice a day
  Soluble Corn Fiber (SCF) without Calcium: Participants consumed a supplement with 12 g/day of SCF for 12 months
- Placebo: This group received a similar supplement without SCF or calcium, administered twice a day
  Placebo: Participants consumed a supplement without SCF or calcium carbonate for 12 months
- Placebo + Calcium: This group received a similar supplement without SCF + 600 mg/d of elemental calcium carbonate, administered twice a day
  Placebo + calcium: Participants consumed a supplement without SCF + calcium carbonate (600 mg/day) for 12 months
Period: Overall Study
Arm/Group | Soluble Corn Fiber (SCF) + Calcium | Soluble Corn Fiber (SCF) Without Calcium | Placebo | Placebo + Calcium
Started | 45 | 43 | 43 | 46
Completed | 40 | 38 | 36 | 37
Not Completed | 5 | 5 | 7 | 9

BASELINE CHARACTERISTICS:
Population: All randomized participants with available baseline data were included in this analysis. Baseline characteristics were assessed prior to study intervention and are summarized by treatment group (Placebo, Placebo + calcium, Soluble Corn Fiber (SCF) without calcium, and Soluble Corn Fiber (SCF) + Calcium).
Groups:
- Total: Total of all reporting groups
Arm/Group | Soluble Corn Fiber (SCF) + Calcium | Soluble Corn Fiber (SCF) Without Calcium | Placebo | Placebo + Calcium | Total
Number analyzed (Participants) | 45 | 43 | 43 | 46 | 177
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.9 (1.35) | 12.1 (1.51) | 12.0 (1.23) | 12.4 (1.4) | 12.1 (1.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 17 | 23 | 20 | 85
  Male | 20 | 26 | 20 | 26 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 32 | 33 | 27 | 128
  Not Hispanic or Latino | 9 | 11 | 10 | 19 | 49
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 1 | 1 | 5
  Asian | 2 | 1 | 1 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 3 | 8 | 5 | 22
  White | 17 | 24 | 15 | 24 | 80
  More than one race | 4 | 0 | 0 | 3 | 7
  Unknown or Not Reported | 13 | 15 | 18 | 11 | 57
Tanner stage [Mean (Standard Deviation); unit: score] — The Tanner Stage is a standardized clinical scale that measures pubertal development based on physical characteristics. It assesses the degree of sexual maturation in children and adolescents by evaluating secondary sexual characteristics such as breast development (in females), genital development (in males), and pubic hair growth (in both sexes). It is rated on a 5-point ordinal scale, with scores ranging from 1 to 5, representing increasing levels of sexual maturity. A higher scores (5) indicate greater pubertal maturation while a lower scores (1) indicate less pubertal maturation.
  score | 2.73 (1.35) | 2.57 (1.24) | 2.74 (1.23) | 2.76 (1.13) | 2.70 (1.23)
Weight [Mean (Standard Deviation); unit: kg] | 46.8 (11.5) | 46.7 (10.6) | 44.6 (12.4) | 47.1 (10.6) | 46.3 (11.2)
Height [Mean (Standard Deviation); unit: cm] | 151.8 (10.8) | 151.8 (11.0) | 149.1 (11.1) | 154.1 (8.36) | 151.7 (10.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Whole Body Bone Mineral Content (BMC)
Description: Participants underwent a bone scan at baseline and after 12-months in the intervention using a dual energy x-ray absorptiometry (DXA)
Time Frame: 12 months
Population: A total of 151 children completed the 12 months visit. Results are presented as change from baseline to the 12 months visit.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Soluble Corn Fiber (SCF) + Calcium | Soluble Corn Fiber (SCF) Without Calcium | Placebo | Placebo + Calcium
Number analyzed (Participants) | 40 | 38 | 36 | 37
grams | 20.1 (11.8) | 18.6 (10.5) | 17.3 (9.2) | 20.7 (10.6)
Statistical Analysis 1: Comparison: Soluble Corn Fiber (SCF) Without Calcium vs Placebo; The main analyses were performed on an intention-to-treat basis. For the primary analysis, percent change from baseline in whole-body BMC after one year of supplement (SCF) vs placebo (AIM 1), we used analysis of covariance, adjusted for baseline age, sex, Tanner stage (puberty status), percent change in weight, and percent change in height. Effects were considered significant at the alpha level of 0.05; Test type: Superiority — Power calculations were done for Aim 1, so the main analysis was done only between SCF and placebo. Significance was set at a p value <0.05; p = 0.377, ANCOVA — We adjusted the models for baseline age, sex, Tanner stage (puberty status), percent change in weight, and percent change in height; We adjusted the models for baseline age, sex, Tanner stage (puberty status), percent change in weight, and percent change in height; Mean Difference (Net) = 1.7, 95% CI 2-sided [-2.12 to 5.53], Standard Error of Mean 1.92
Statistical Analysis 2: Comparison: Soluble Corn Fiber (SCF) + Calcium vs Placebo + Calcium; The main analyses were performed on an intention-to-treat basis. For the secondary analysis, percent change from baseline in whole-body BMC after one year of supplement (SCF+calcium) vs placebo+calcium (AIM 2), we used analysis of covariance, adjusted for baseline age, sex, Tanner stage (puberty status), percent change in weight, and percent change in height. Effects were considered significant at the alpha level of 0.05; Test type: Superiority — Significance was set at a p value <0.05; p = 0.245, ANCOVA; Mean Difference (Net) = 1.950, 95% CI 2-sided [-1.366 to 5.266], Standard Deviation 1.8

2. Secondary Outcome: Change in Spine BMC
Description: as for outcome 1
Time Frame: 12 months
Population: A total of 151 children completed the 12 months visit, but data from 1 child in the placebo+calcium group for BMC lumbar spine was not included as the DXA machine gave an error and it was not resolved in time and the child did not come back. Results are presented as change from baseline to the 12 months visit.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Soluble Corn Fiber (SCF) + Calcium | Soluble Corn Fiber (SCF) Without Calcium | Placebo | Placebo + Calcium
Number analyzed (Participants) | 40 | 38 | 36 | 36
grams | 21.8 (14.5) | 18.7 (10.8) | 22.4 (13.2) | 23.8 (16.1)
Statistical Analysis 1: Comparison: Soluble Corn Fiber (SCF) Without Calcium vs Placebo; The main analyses were performed on an intention-to-treat basis. For the secondary analysis, percent change from baseline in lumbar BMC after one year of supplement (SCF) vs placebo, we used analysis of covariance, adjusted for baseline age, sex, Tanner stage (puberty status), percent change in weight, and percent change in height. Effects were considered significant at the alpha level of 0.05; Test type: Superiority; p = 0.05, ANCOVA; Mean Difference (Net) = 1.655, 95% CI 2-sided [-0.765 to 8.143]
Statistical Analysis 2: Comparison: Soluble Corn Fiber (SCF) + Calcium vs Placebo + Calcium; Test type: Superiority; p = 0.05, ANCOVA; Mean Difference (Net) = 1.035, 95% CI 2-sided [-7.680 to 2.435], Standard Error of Mean 2.535

ADVERSE EVENTS:
Time Frame: 1 year
Description: Serum calcium
Arm/Group | Soluble Corn Fiber (SCF) + Calcium | Soluble Corn Fiber (SCF) Without Calcium | Placebo | Placebo + Calcium
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/43 | 0/43 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/43 | 0/43 | 0/46
Other Adverse Events (participants affected / at risk) | 3/45 | 1/43 | 0/43 | 3/46
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Soluble Corn Fiber (SCF) + Calcium (N=45) | Soluble Corn Fiber (SCF) Without Calcium (N=43) | Placebo (N=43) | Placebo + Calcium (N=46)
Gastrointestinal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Low bone mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
High serum calcium (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-26): https://cdn.clinicaltrials.gov/large-docs/62/NCT02916862/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-24): https://cdn.clinicaltrials.gov/large-docs/62/NCT02916862/ICF_001.pdf